CLINICAL TRIAL: NCT01289392
Title: Effects of the Treatment With Continuous Positive Airway Pressure (CPAP) and Oral Appliance, Associated or Not Associated With Physical Exercise, in the Obstructive Sleep Apnea
Brief Title: Continuous Positive Airway Pressure (CPAP), Oral Appliance and Physical Exercise in the Obstructive Sleep Apnea
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Associação Fundo de Incentivo à Pesquisa (Other)
Responsible Party: Principal Investigator, Prof. Dr. Lia Azeredo-Bittencourt, professor, Associação Fundo de Incentivo à Pesquisa
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: CEP 0352/09
Record Dates: First submitted 2011-01-31; First posted 2011-02-03 (Estimated); Results first posted 2013-04-12 (Estimated); Last update posted 2013-05-03 (Estimated); Status verified 2013-03

CONDITIONS: Obstructive Sleep Apnea
Keywords: Obstructive Sleep Apnea; CPAP; Oral appliance; Aerobic exercise; Resistance training
MeSH Terms: conditions — Sleep Apnea, Obstructive | interventions — Continuous Positive Airway Pressure; Exercise

STUDY DESIGN:
Who Masked: Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (3):
- Continuous Positive Airway Pressure (CPAP) (Active Comparator): CPAP is the gold standard treatment
  Interventions: Device: Continuous Positive Airway Pressure (CPAP)
- Oral Appliance (Active Comparator): Alternative treatment for obstructive sleep apnea patients
  Interventions: Device: Oral Appliance (OA)
- Physical Exercise (Active Comparator): Aerobic and resistance physical exercises
  Interventions: Behavioral: Physical Exercise

INTERVENTIONS:
Device: Continuous Positive Airway Pressure (CPAP) — Previously determinated airway pressure: used for two months unassociated with physical exercise and used for four months associated with physical exercise
  Arms: Continuous Positive Airway Pressure (CPAP)
Device: Oral Appliance (OA) — Anterior mandibular repositioner: used for two months unassociated with physical exercise and used for four months associated with physical exercise
  Arms: Oral Appliance
Behavioral: Physical Exercise — aerobic and resistance Physical exercise, three times a week, for four months
  Arms: Physical Exercise

SUMMARY:
Introduction: It is unclear whether exercise training with or without Continuous Positive Airway Pressure (CPAP) and Oral Appliance (OA) is more effective in reducing symptoms of Obstructive Sleep Apnea (OSA) than treatment solely with CPAP or OA.

Objective: In patients with moderate OSA, the investigators will evaluate the effect on the subjective and objective measures of sleep, quality of life and mood of different forms of treatment: exercise training of 4 months; exercise training of 4 months associated with CPAP and OA; treatment with CPAP and treatment with OA.

Material and Methods: Sixty male patients (25-65 years, sedentary lifestyle, Body Mass Index (BMI) < 35kg/m2, Apnea-Hypopnea Index (AHI) between 15-30/h, Epworth sleepiness scale > 9) will be divided into three groups: CPAP+exercise group (CE; n=20), OA+exercise group (AE; n=20), and Exercise training group (E; n=20). The patients in groups CE and AE will complete two months of treatment with CPAP or OA to examine the separate effects of these devices. As the patients of the E group did not use the CPAP but will undergo four months of exercise training. After this initial step, patients in CE and AE groups will undergo four months of exercise training associated with CPAP or OA. The investigators will evaluate the subjective sleep parameters (sleep disorders questionnaire, the Epworth Sleepiness Scale, sleep diaries) and objective (polysomnography), Short Form Health Survey (SF-36), Questionnaire Profile of Mood States (POMS) and anthropometric measurements (neck circumference and body composition), the incremental exercise test (ergospirometry) and the one Repetition Maximum test (1RM).

ELIGIBILITY:
Inclusion Criteria:

* Male subjects aged between 25 and 65 years old
* Sedentary according to the criteria of Godin and Shephard (1985) and / or ACSM (2000)
* Epworth Sleepiness Scale over score of nine
* Normal range of laboratory tests [blood count, cholesterol, High-density lipoprotein (HDL), triglycerides, fasting glucose, creatinine, Thyroid-stimulating hormone (TSH)]
* Lung function test (spirometry), chest X-ray (for smokers and former smokers) electrocardiogram (rest and stress) and ENT examination without significant changes

Exclusion Criteria:

* Presence of clinical diseases (chronic obstructive pulmonary disease, asthma, interstitial lung diseases, neuromuscular diseases, heart failure, thyroid disease, rheumatologic and psychiatric) and other sleep disorders
* Presence of anatomical obstructive upper airway, tonsil grade III and IV septal deviation and grade III (severe) that may affect the outcome of CPAP
* Loss of posterior dental support to undermine the retention of oral appliance
* Active periodontal disease, compared Dental crown / dental root less than or equal to 1 (c / r ≤ 1), need for primary dental care (cavities, root canal treatment or retreatment, dentures, ie outlying), open bite
* Protrusive displacement less than five millimeters
* Limited mouth opening (would prevent the forming of the dental arches)
* Alcoholism
* Uuse of sleep-inducing medications
* Habits or occupations that lead to sleep deprivation or alteration of the sleep-wake cycle
* Inability to perform physical exercise, regular history sports activities
* Intolerance to Continuous Positive Airway Pressure (CPAP)
* Obesity grade II (moderate) and III (severe)

Ages: 25 Years to 65 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 25 (Actual)
Dates: Start 2010-10; Primary Completion 2013-01 (Actual)

CONTACTS AND LOCATIONS:
Locations (1):
- Instituto do Sono/Associação Fundo de Incentivo a Psicofarmacologia, São Paulo, São Paulo, Brazil

REFERENCES:
- [Derived] Schutz TC, Cunha TC, Moura-Guimaraes T, Luz GP, Ackel-D'Elia C, Alves Eda S, Pantiga G Jr, Mello MT, Tufik S, Bittencourt L. Comparison of the effects of continuous positive airway pressure, oral appliance and exercise training in obstructive sleep apnea syndrome. Clinics (Sao Paulo). 2013;68(8):1168-74. doi: 10.6061/clinics/2013(08)17. PMID 24037015

RESULTS

PARTICIPANT FLOW:
Recruitment Details: sleep disorder clinic
Groups:
- Continuous Positive Airway Pressure (CPAP): CPAP is the gold standard treatment
  Continuous Positive Airway Pressure (CPAP) : Previously determinated airway pressure: used for two months unassociated with physical exercise and used for four months associated with physical exercise
- Oral Appliance: Alternative treatment for obstructive sleep apnea patients
  Oral Appliance (OA) : Anterior mandibular repositioner: used for two months unassociated with physical exercise and used for four months associated with physical exercise
- Physical Exercise: Aerobic and resistance physical exercises
  Physical Exercise : aerobic and resistance Physical exercise, three times a week, for four months
Period: Overall Study
Arm/Group | Continuous Positive Airway Pressure (CPAP) | Oral Appliance | Physical Exercise
Started | 9 | 9 | 7
Completed | 9 | 9 | 7
Not Completed | 0 | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Continuous Positive Airway Pressure (CPAP) | Oral Appliance | Physical Exercise | Total
Number analyzed (Participants) | 9 | 9 | 7 | 25
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0 | 0
  Between 18 and 65 years | 9 | 9 | 7 | 25
  >=65 years | 0 | 0 | 0 | 0
Age Continuous [Mean (Standard Deviation); unit: years] | 38.62 (8.15) | 42.33 (6.20) | 42.28 (8.28) | 41.10 (7.27)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 0 | 0 | 0 | 0
  Male | 9 | 9 | 7 | 25
Region of Enrollment [Number; unit: participants]
  Brazil | 9 | 9 | 7 | 25

OUTCOME MEASURES:

1. Primary Outcome: Objective Sleep Parameters
Description: Polysomnographic date of sleep stages percentages, sleep efficiency, arousals, apnea-hypopnea index, oxyhemoglobin saturation
Time Frame: 6 months after the basal evaluation
Reporting Status: Not Posted

2. Secondary Outcome: Inflammatory Markers
Description: Blood samples to test: tumor necrosis factor-alpha (TNF-alpha), C-reactive protein (CRP), Interleukin-6 and Interleukin-8
Time Frame: 6 months after the basal evaluation
Reporting Status: Not Posted

3. Primary Outcome: Sleep Apnea
Description: Number of events per hour of sleep
Time Frame: 6 months
Measure: Mean (Standard Deviation); unit: number of events
Arm/Group | Continuous Positive Airway Pressure (CPAP) | Oral Appliance | Physical Exercise
Number analyzed (Participants) | 9 | 9 | 7
number of events | 25.06 (10.54) | 30.76 (19.00) | 22.81 (12.77)

ADVERSE EVENTS:
Arm/Group | Continuous Positive Airway Pressure (CPAP) | Oral Appliance | Physical Exercise
Serious Adverse Events (participants affected / at risk) | 0/9 | 0/9 | 0/7
Other Adverse Events (participants affected / at risk) | 0/0 | 0/0 | 0/0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No